CLINICAL TRIAL: NCT00787098
Title: Investigating Modes of Progressive Mobility
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hill-Rom (Industry)
Responsible Party: Chris Winkelman, RN, PhD, Assistant Professor, Case Western Reserve University, Francis Payne Bolton School of Nursing
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR-0076
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2009-07-03 (Estimated); Status verified 2009-07

CONDITIONS: Critical Care; Mechanical Ventilation; Intensive Care; Muscular Atrophy
Keywords: therapeutic mobility; acute care; nursing; inflammatory markers
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): RA begins data collection with chart review for demographic and explanatory variables, collects data for baseline muscle strength. During standard care period, PM will obtain information about the plan for activity for enrolled patients (turning, complete or partial weight-bearing i.e., reverse Trendelenberg positioning, ROM, sitting and walking) through discussion with the direct providers. RA will interview one provider about factors which influence the decision to implement activity or provide bedrest, including the presence of orders for bedrest or physical therapy. If activity is planned, the PM will observe and record the type and duration of activity, drawing serum biomarkers 20 minutes before and 20 minutes after the activity. If no activity is planned or activity duration is less than 10 minutes, serum for only baseline inflammatory biomarkers will be drawn. The RA will collect outcomes data within 24 hours of discharge from the ICU.
- 2 (Experimental): Identical procedures for date recruitment, consent and data collection will occur. In this phase, the Project Manager will promote the use of the ETM protocol through coaching (e.g., reminding staff of benefits of mobility, identification of available resources, or suggesting cessation of bedrest orders) and by participating in planning at least one 20-minute activity.
  Interventions: Other: ETM protocol

INTERVENTIONS:
Other: ETM protocol — ETM is 4 levels. Level 1, each receives repositioning from lateral to supine positions at even hours, totaling 60 minutes of activity/positioning over 24 hours. If tolerated, two periods of 20 minutes of supine position with a reverse trendelenberg position of 15-20 degrees will be used to promote orthostasis. Level 2 is turning every 2 hours, positioning in reverse trendelenberg at 15-25 degrees as tolerated, active resistance with ICU staff for 20 minutes daily for a total of 60-80 minutes of activity/positioning daily. At Level 3, 2 times 20 minutes of a sitting are added to active ROM and inbed turning (estimated 80-100 total minutes of activity daily). Sitting is in bed or with non-weightbearing assisted transfer to chair with backrest elevation at 75-90 degrees and legs in a dependent position. Level 3 interventions; minimal weight-bearing. Level 4, weight-bearing transfer to chair and ambulation are added to inbed turning.
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effects of specific activities with and without an early therapeutic mobility (ETM) protocol among patients who experience three or more days of mechanical ventilation. A second purpose is to examine staff/delivery system and patient factors that influence the initiation and progression of activity with and without an ETM protocol. The hypothesis is that ETM protocols will result in improved patient outcomes.

DETAILED DESCRIPTION:
The specific aims of this study are to:

1. Compare patient responses to selected modes of therapy (activity) without and with an ETM protocol

   1. Molecular responses: markers of inflammation interleukin (IL)-6 and IL-10
   2. Physiological responses: peripheral oxygen saturation, heart rate, blood pressure, new dysrhythmias
   3. Safety/Unsafe events including pain, fatigue, line or tube dislodgement, fall or near fall
2. Determine the associations between duration and level of activity/ETM achieved and outcomes:

   1. occurrence of delirium
   2. occurrence of ventilator associated pneumonia
   3. occurrence of deep vein thrombosis or pulmonary emboli
   4. occurrence of acquired pressure ulcer
   5. muscle strength
   6. number of days mechanically ventilated
   7. discharge location (after ICU)
3. Describe strategies used in the ICU to initiate and implement activity with and without an ETM protocol

   1. use of personnel such as registered nurses, physical therapists, respiratory therapist and nursing assistants
   2. use of equipment such as a walker, lift device, belt or bed
   3. perception of sufficient time and abilities
4. Describe patient factors that are associated with implementation of ETM

   1. Potentially modifiable exemplars: sedation, site of vascular access, physician orders
   2. Potentially nonmodifiable exemplars: weight, consciousness, hemodynamic instability, terminal condition

This is a prospective, longitudinal, repeated measures study with a control period, run-in period and intervention period. Data will be collected during all three periods for comparison. During the control period, patients will receive standard care. Standard care in this institution does not include a program of progressive or early mobility but does include activities similar to the ETM protocol, implemented at the discretion of the staff. During the run-in period, subjects will receive a mix of standard care and the intervention.

ELIGIBILITY:
Inclusion Criteria:

* P:F ratio > 100
* FiO2 < 60% and PEEP less than 10 cmH20
* hemodynamic stability ten minutes after turning (i.e., heart rate (HR) and/or systolic blood pressure (BP) changes less than 20% of baseline)
* baseline (rest) vitals signs of HR 50-110
* mean arterial pressure (MAP) 60-100 mmHg
* peripheral oxygenation saturation (SpO2) greater than 88%
* Sufficient cognition for progression to levels 2-4 of ETM to assist with out of bed positioning or movement
* a high degree of dependency on others for positioning is acceptable
* there are no exclusions based on gender or minority status.

Exclusion Criteria:

* End-stage muscular dystrophy
* myasthenia gravis
* new quadriplegia
* coma
* increased intracranial pressure
* unrepaired hip fracture and multiple lower extremity fractures
* Patients experiencing active titration of intravenous vasoactive medications (e.g. dopamine, epinephrine, or norepinepherine) will be excluded
* concurrent use of a continuous lateral rotation bed
* patients for high risk of death will also be excluded
* MICU admission following a hospital stay of >9 days in the past months
* age >80 in the presence of 2 or more life-threatening illnesses
* diagnosis of an active stage IV malignancy
* status post cardiac arrest
* diagnosis of intracerebral hemorrhage requiring mechanical ventilation
* subjects over 400 pounds can be excluded from mobilization based on the judgment of the bedside nurse or project manager; if the risk for staff or patient harm from moving a patient with excessive weight is considered likely, mobilization will not occur.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Compare immediate molecular and physiological patient responses to activity with responses to an ETM protocol. | 1, 2, 3, 7, days then weekly

SECONDARY OUTCOMES:
A secondary aim is to identify strategies and conditions that promote or prevent ETM. | 1, 3, 5, 7, days then weekly

CONTACTS AND LOCATIONS:
Overall Officials: Chris Winkelman, PhD, Principal Investigator — Case Western Reserve University

REFERENCES:
- [Background] Morris PE, Goad A, Thompson C, Taylor K, Harry B, Passmore L, Ross A, Anderson L, Baker S, Sanchez M, Penley L, Howard A, Dixon L, Leach S, Small R, Hite RD, Haponik E. Early intensive care unit mobility therapy in the treatment of acute respiratory failure. Crit Care Med. 2008 Aug;36(8):2238-43. doi: 10.1097/CCM.0b013e318180b90e. PMID 18596631